CLINICAL TRIAL: NCT01121211
Title: Hormonal Factors in the Treatment of Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009P-001845/1; 5R01MH083657-05A2 (NIH)
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Anorexia Nervosa; Eating Disorder; Anxiety; Depression
Keywords: Testosterone; Hormones; Mental Health
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Anxiety Disorders; Depression; Psychological Well-Being | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone (Active Comparator): Testosterone x 24 weeks
  Interventions: Drug: Testosterone
- Placebo (Placebo Comparator): Placebo x 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone — Testosterone 300mcg transdermal patch x 24 weeks.
  Arms: Testosterone
Drug: Placebo — Placebo transdermal patch x 24 weeks
  Arms: Placebo

SUMMARY:
The investigators are investigating whether a hormone that is naturally produced by the human body, called testosterone, can help improve weight, disordered eating, depression, and anxiety. The investigators hypothesize that testosterone will be a novel and effective endocrine-targeted therapy for patients with anorexia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 45 years; if participating in the neuroimaging sub study, age 18-40
* Meet DSM-IV criteria for AN (restricting or binge/purge type, BMI 15-17.5) OR meet criteria for sub-threshold AN, i.e., all DSM-IV criteria except that patients can have a BMI of <18.5 kg/m2 with or without amenorrhea.
* Free T below the median for healthy women of reproductive age
* All participants will be required to have a treatment team in place that consists of (at least) a primary care physician and a psychotherapist. Participants will need to have had regular contact with a primary care physician and be in an individual psychotherapy program. Participants will agree to continue with this treatment team and therapy throughout the active course of the study. If participants are taking psychotropic medications, the dose must be stable for 3 months before study entry

Exclusion Criteria:

* Pregnant women or women of child bearing potential who are not using medically accepted means of contraception (to include oral contraceptive, patch or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy).
* Unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic
* Serious suicide risk, substance use disorder active within last 6 months, bipolar I disorder, severe current depressive symptoms (indexed by HAM-D score >20 [excluding 2 eating/weight loss items related to the symptoms of AN]), or psychotic disorder
* New psychotropic drug regimen, specifically a significant dose change or change in drug class, within the last 6 weeks. A study psychiatrist will assess whether PRN medications and dose changes are clinically significant enough to defer enrollment of specific potential study subjects.
* Untreated hypothyroidism
* If receiving estrogen therapy, including oral contraceptives or transdermal estrogen therapy, significant change in dose in the prior 3 months
* Use of androgens or androgen precursors, including T, DHEA and methyl T, within 3 months
* Any investigational psychotropic drug within the last 3 months
* In the judgment of the study clinician, unlikely to be able to participate safely throughout the study period
* Alanine aminotransferase (ALT) > 2x upper limit of normal
* Creatinine >1.5x upper limit
* Serum potassium < lower limit of normal
* If participating in the sub study, unable to tolerate 1 hour in MRI; contraindication to MRI (such as implanted pacemaker, cerebral aneurysm clips, extensive orthopedic hardware instrumentation); gastrointestinal tract surgery (including gastrectomy, gastric bypass surgery, and small or large bowel resection); history of psychosis by SCID

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — Massachusetts General Hospital; Karen K Miller, MD, Study Director — Massachusetts General Hospital; Erinne Meenaghan, NP, Study Chair — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Plessow F, Galbiati F, Eddy KT, Misra M, Miller KK, Klibanski A, Aulinas A, Lawson EA. Low oxytocin levels are broadly associated with more pronounced psychopathology in anorexia nervosa with primarily restricting but not binge/purge eating behavior. Front Endocrinol (Lausanne). 2023 Jan 31;13:1049541. doi: 10.3389/fendo.2022.1049541. eCollection 2022. PMID 36798485
- [Derived] Kimball A, Schorr M, Meenaghan E, Bachmann KN, Eddy KT, Misra M, Lawson EA, Kreiger-Benson E, Herzog DB, Koman S, Keane RJ, Ebrahimi S, Schoenfeld D, Klibanski A, Miller KK. A Randomized Placebo-Controlled Trial of Low-Dose Testosterone Therapy in Women With Anorexia Nervosa. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4347-4355. doi: 10.1210/jc.2019-00828. PMID 31219558

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone | Placebo
Started | 43 | 47
Completed | 32 | 35
Not Completed | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Testosterone: Testosterone x 24 weeks
  Testosterone: Testosterone 300mcg transdermal patch x 24 weeks.
  Placebo: Placebo transdermal patch x 24 weeks
- Placebo: Placebo x 24 weeks
  Testosterone: Testosterone 300mcg transdermal patch x 24 weeks.
  Placebo: Placebo transdermal patch x 24 weeks
- Total: Total of all reporting groups
Arm/Group | Testosterone | Placebo | Total
Number analyzed (Participants) | 43 | 47 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 47 | 90
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7) | 27 (7) | 27 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 47 | 90
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 47 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight
Description: Weight in kilograms
Time Frame: Baseline, 24 Weeks
Population: All subjects who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 42 | 46
kilograms | 0.1 (2.7) | 1.5 (3.2)

2. Primary Outcome: Change From Baseline in Depression Symptom Severity
Description: Hamilton Depression Rating Scale (HAM-D) (Higher score = greater depression symptom severity; Score Range 0 - ≥ 23)
Time Frame: Baseline, 24 weeks
Population: All subjects who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: HAM-D score on a scale
Arm/Group | Testosterone | Placebo
Number analyzed (Participants) | 42 | 46
HAM-D score on a scale | -3 (5) | -3 (5)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Testosterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/47
Serious Adverse Events (participants affected / at risk) | 4/43 | 1/47
Other Adverse Events (participants affected / at risk) | 33/43 | 33/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=43) | Placebo (N=47)
Hospitalization due to anorexia nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization due to exacerbation of GI disorders (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospitalization due to depression exacerbation (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone (N=43) | Placebo (N=47)
Acne or Increase in acne (Skin and subcutaneous tissue disorders) | 14 (24) | 18 (24) — Adverse event data collected at each study visit.
Patch site irritation (Skin and subcutaneous tissue disorders) | 12 (12) | 15 (15) — Adverse event data collected at each study visit.
Oily skin or Increase in oily skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) — Adverse event data collected at each study visit.
Hirsutism or Increased hair growth (Skin and subcutaneous tissue disorders) | 9 (15) | 10 (15) — Adverse event data collected at each study visit.
Depilation (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) — Adverse event data collected at each study visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes